CLINICAL TRIAL: NCT04259177
Title: Turkish Validity And Reliability Of The Hammersmith Infant Neurological Evaluation (Hine)
Acronym: Hine
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adıgüzel, Msc PhD. cd. Lecturer, Sanko University
Other Study IDs: SankoUnv
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy; Reliability; Infant Development; Infant, Premature, Diseases; Infant Asphyxia; Validity
Keywords: Reliability; Validity; Hammersmith Infant Neurological Evaluation (HINE); Turkish version; Infant
MeSH Terms: conditions — Cerebral Palsy; Infant, Premature, Diseases | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Scale — This test is divided into 3 sections: neurological examination, developmental motor boundary stones and behavioral status, and consists of a total of 37 items. The first part consists of 26 items such as cranial nerve functions, posture, quality, amount of movements, muscle tone, reflex and reactions. The second part evaluates motor development boundary stones consisting of 8 items. The third part refers to the behavioral condition consisting of 3 items. These items can be easily scored. It can be rated as optimal or inadequate. Each item is scored separately (as 0, 1, 2, 3) and the final total score is calculated. The total score ranges from 0-78. The total score shows the global optimal scores.
  Other Names: evaluation

SUMMARY:
The high risk of infants are defined as having a negative environmental and biological factor history, where these factors can lead to neuromotor development problems. It is a heterogeneous group of premature babies born under the age of thirty-seven weeks, with a low birth weight term or infants with developmental retardation due to various reasons. Risk factors in preterm infants include perinatal asphyxia, hypoxic ischemic encephalopathy (HIE), periventricular leukomalacia (PVL), intraventricular hemorrhage (IVH), respiratory distress syndrome (RDS), broncho pulmonary dysplasia (BPD), hyperbilirubinemia, infection. alcohol syndrome, muscle tone disorders, low birth weight, hydrocephalus and microcephaly. These babies, especially preterm infants with low birth weight, may encounter a neurological sequence such as Cerebral Palsy (CP), epilepsy, hearing and vision loss, mental retardation, language-speech, behavioral problems and learning difficulties. CP is the most common disease of childhood, with the possibility of occurrence in 2-3 / 1000 live births.Today, the effectiveness of various methods has been proven to make early diagnosis of CP. One of these methods is the Hammersmith Infant Neurological Evaluation (HINE).

DETAILED DESCRIPTION:
The diagnosis of CP, which can be observed with high risk infants, is based on the observation of many neurological and clinical signs. The diagnosis usually takes place between 12-24 months. In the past years, before 12-24 months, it was seen as a hidden or silent period that could not be fully defined in terms of CP. However, today this definition has been found invalid because the diagnosis of 'high risk of CP' or CP can be predicted precisely before the corrected 6 months.There are 3 methods with the best predictable validity of determining CP before the corrected 5-month period: Neonatal Magnetic Resonance Imaging (MRI) (86% -89% sensitivity), Prechtl's Qualitative General Movement Assessment (GMs) (98% sensitivity), Hammersmith Infant Neurological Evaluation (HINE) (90% sensitivity). Various difficulties are encountered in long-term follow-up of infants who are discharged from neonatal intensive care units (NICU) in developing countries. Many of these infants are referred to pediatricians or pediatric neurologists as needed. Others are not routinely monitored. However, in order to encourage more consistent and disciplined early assessments for high-risk infants, the guides applied should be adapted to neonatal follow-up clinics. For this reason, various health professionals working in the field of Pediatrics should be supported in providing objective tests and training materials in order to provide coordination and create a common language in the follow-up process. It is known that the HINE test does not require certification training and whose reliability is valid, does not have a Turkish version. Using proven methods to determine these needs and to direct the necessary professionals is a more important guide for clinicians. In order to meet the needs in this field, the Turkish version of the HINE scale in 6-12 months of infants was adapted and this validity and reliability study was planned.

ELIGIBILITY:
Inclusion Criteria:

* Infants with periventricular hemorage, intracranial hemorage,grade 2, 3, 4, cystic periventricular leukomalacia, stage 3 hypoxic ischemic encephalopathy, neonatal bilirubin encephalopathy (kernicterius), perinatal stroke, perinatal asphyxia, hydrocephalus
* Chronic lung disease, respiratory lung disease (RDS), broncho pulmonary dysplasia and babies with long-term o₂ support
* Gram negative bacterial sepsis, necrotizing enterocolitis (NEC), infantile apnea, preterm babies with cerebral malformation
* Low Apgar score (3 and below), Preterm babies with intrauterine growth retardation, multiple births (twins, triplets), Premature Retinopathy (ROP)
* Infants with prolonged severe hypoglycaemia and hypocalcemia
* Surgical conditions such as diaphragmatic hernia or tracheoesophageal fistula
* Infants who are small for gestational age (small for gestational age, sga, less than 3rd percentile) or large for gestational age (large for gestational age, LGA, greater than 97th percentile)
* Infants who received mechanical ventilation for more than 24 hours
* Infants younger than 32 gestational weeks and under 1500 kilograms

Exclusion Criteria:

* Infants with congenitalmal formation (spina bifida, congenital muscular torticollis, arthrogryposis multiplex congenita..vs)
* Infants diagnosed with metabolic and genetic diseases (down syndrome, spinal muscular atrophy, duchenne muscular dystrophy..vs)
* Postterm Infants still dependent on intubation and mechanical ventilator at 3 months.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Infants with high risk of cerebral palsy (CP) with the age of 3-12 months.
  * Infants with healthy peers of high of cerebral palsy infants.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
magnetic resonance imaging (MRI) | first day of assessment
  magnetic resonnas imaging method is an imaging method that shows the parts of the brain that are damaged without oxygen. Imaging is obtained by sending rays to the brain with sound waves.
Prechtl's general movements (GMs) analysis | up to 5 months
  Gms can identify neurological issues predictive of cerebral palsy and other developmental disabilities.GMs videos around 3 months of age (12-16 weeks corrected age) provide the most predictive information about the likelihood risk of cerebral palsy. Ther isn't maximum or cut off scores.Movements are noted as observed/or not. Also quality of fidgety movements are scored as low or high quality.

SECONDARY OUTCOMES:
prenatal,natal and postnatal risk factors | up to 1 year
  These parameter can be the risk of Cerebral Palsy for infants. Infants with periventricular bleeding, intracranial bleeding grade 2, 3, 4, cystic periventricular leukomalacia, stage 3 hypoxic ischemic encephalopathy, neonatal bilirubin encephalopathy (kernicterius), perinatal stroke, perinatal asphyxia, hydrocephalus.Chronic lung disease, respiratory lung disease (RSD), broncho pulmonary dysplasia and babies with long-term o₂ support Gram negative bacterial sepsis, necrotizing enterocolitis (NEC), preterm babies with cerebral malformation. Low Apgar score (3 and below), Preterm babies with intrauterine growth retardation, multiple births, Premature Retinopathy (ROP). Babies with prolonged severe hypoglycaemia and hypocalcemia. Infants who are small for gestational age or large for gestational age. Infants who received mechanical ventilation for more than 24 hours. Babies younger than 32 gestational weeks and under 1500 kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD cd., Principal Investigator — sanko Üniversitesi
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided